CLINICAL TRIAL: NCT04988438
Title: Gastrointestinal Motor Disorders (Esophageal and Anorectal) in Patients After COVID-19 Infection
Brief Title: Gastrointestinal Motor Disorders (Esophageal and Anorectal) After COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Žarko Babić, Principal investigator, Clinical professor, Heat of Interventional gastroenterology, University Hospital Dubrava
Other Study IDs: 2021/1407-03UHD
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Motility Disorder
Keywords: After COVID-19; gastrointestinal motility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- esophageal manometry: The patients who has previously mentioned symptoms will underwent to manometry monitoring of esophageal and anorectal disorders.
  For this investigation we have proven normal and standardized manometric values on previous investigations by other authors, so the control group is not needed. We know the normal manometric values (Chicago 3 score).
- anorectal manometry: The patients who has previously mentioned symptoms will underwent to manometry monitoring of esophageal and anorectal disorders.
  For this investigation we have proven normal and standardized manometric values on previous investigations by other authors, so the control group is not needed. We know the normal manometric values (London protocol).

SUMMARY:
The patients who had COVID-19 infection, and after that reported for one of the signs of gastrointestinal disorder (esophageal and anorectal) will be underwent to esophageal and anorectal motor monitoring investigation (HRM manometry) on standard protocol.

DETAILED DESCRIPTION:
The patients who had COVID-19 infection, and after that reported for one of the signs of gastrointestinal (esophageal and anorectal disorder) will be underwent to esophageal and anorectal motor monitoring investigation (HRM manometry) on standard protocol.

The patients with dysphagia, chest discomfort during swallowing, or chest pain during swallowing, patients with obstipation, fecal evacuation symptoms, lower stomach discomfort before defecation etc. will be included in the study. In all of them other gastrointestinal diseases will be excluded by standard routine laboratory investigation, ultrasound, routine endoscopy investigation and 24 hours impedance pH-measurement.

After manometric measurement of esophagus and anorectal region to standard protocol by using MMS-HRM 360 monitoring system with 36 canals catheter for esophagus and 24 canals catheter for anorectal monitoring, data will be calculated by using statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal and anorectal symptoms after COVID 19- infection
* Patients with worsening of esophageal and anorectal symptom after COVID 19- infection, but who had previously described esophageal and anorectal symptoms

Exclusion Criteria:

* Other gastrointestinal disease that can influence to results
* Gastroesophageal reflux
* H. Pylori infection
* Bacterial, parasitic, viral and fungal gastrointestinal infection or infestation
* Myasthenia
* Scleroderma
* Diabetes mellitus
* Thyroidal hyperfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients from 20-80 years, men and women.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of esophageal parameters 1 on manometry | 120 days
  In esophagus we will measure Upper and lower esophageal sphincter pressure in mmHg.
Measurement of esophageal parameters 2 on manometry | 120 days
  In esophagus we will measure Integrated relaxation pressure (IRP) in mmHg.
Measurement of esophageal parameters 3 on manometry | 120 days
  In esophagus we will measure Contractile front velocity (CVF) in cm/s.
Measurement of esophageal parameters 4 on manometry | 120 days
  In esophagus we will measure Distal contractile integral (DCI) in mmHg.s.cm.
Measurement of esophageal parameters 5 on manometry | 120 days
  In esophagus we will measure Distal latency (DL) in seconds.
Measurement of esophageal parameters 6 on manometry | 120 days
  In esophagus we will measure Peristaltic brake (BR) in cm.
Measurement of anorectal parameters 1 on manometry | 2 years
  On anorectal manometry we will measure Resting test pressure in mmHg.
Measurement of anorectal parameters 2 on manometry | 2 years
  On anorectal manometry we will measure Squeeze test pressure in mmHg.
Measurement of anorectal parameters 3 on manometry | 2 years
  On anorectal manometry we will measure Endurance squeeze test pressure in mmHg.
Measurement of anorectal parameters 4 on manometry | 2 years
  On anorectal manometry we will measure recto-anal inhibitory reflex test (RAIR)- relaxation in percent.
Measurement of anorectal parameters 5 on manometry | 2 years
  On anorectal manometry we will measure Push test pressure in mmHg.
Measurement of anorectal parameters 6 on manometry | 2 years
  On anorectal manometry we will measure Sensation test with ml in balloon.
Measurement of anorectal parameters 7 on manometry | 2 years
  On anorectal manometry we will measure Balloon expulsion test as positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Žarko B Babić, prof.dr.sc., Principal Investigator — Head od Interventional gastroenterology UH Dubrava
Locations (1):
- Prof.dr.sc. Žarko Babić, FEBGH, Zagreb, Select State, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Babic Z, Bezdrov L, Haber VE, Kardum D, Andabak M, Rob Z, Banic M. Esophageal motility disorders after COVID-19 infection. Sci Rep. 2025 Dec 6;16(1):1428. doi: 10.1038/s41598-025-31067-1. PMID 41353487